CLINICAL TRIAL: NCT05967390
Title: Localized Analysis of Normalized Distance From Scalp to Cortex and Personalized Evaluation (LANDSCAPE): A Project of MRI-informed Computational Head Model
Brief Title: Localized Analysis of Normalized Distance From Scalp to Cortex and Personalized Evaluation (LANDSCAPE)
Status: Enrolling by invitation | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, LU Hanna, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2018.077; 2018.077 (Other: The Chinese University of Hong Kong)
Record Dates: First submitted 2023-06-15; First posted 2023-08-01 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Aging; Dementia Alzheimers; Parkinson Disease; Dementia Frontotemporal; Depression in Old Age
Keywords: Aging; Scalp-to-cortex distance; Transcranial brain stimulation; Parkinson disease; Simulation; Predictor
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Pick Disease of the Brain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Neurocognitive disorder (NCD): The NCD patients are defined with a chronological age over 60 years and a Montreal Cognitive Assessment (MoCA) total score between 22 and 26.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — One time for each day, lasting for three weeks.

SUMMARY:
Scalp to cortex distance (SCD), as a key technological parameter of brain stimulation, has been highlighted in the guidelines of non-invasive brain stimulation. However, in the context of age-related brain changes, the region-specific SCD and its impact on stimulation-induced electric field in different types of neurodegenerative diseases remain unclear.

DETAILED DESCRIPTION:
Objective: This study aimed to investigate the region-specific SCD and its relationship with morphometric features and cognitive function in age- and disease-specific populations. Methods: The SCD and cortical thickness (CT) of left primary motor cortex (M1) and dorsolateral prefrontal cortex (DLPFC) were measured in cognitively normal adults and dementia patients. CT-adjusted SCD was used to control the influence of CT on SCD. Head model was developed to simulate the impact of SCD on the electric field induced by transcranial electrical stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed as assessed by the Edinburgh Inventory
* Able to attend TMS interventions
* Consent
* Independent in daily life activities

Exclusion Criteria:

* Uncorrected visual or auditive deficits not allowing the realization of the test
* Evolutive disease (such as cancer)
* Neurological or psychiatric antecedent
* Counter-indication to MRI

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy normal ageing adults and adults with neurocognitive disorders
Sampling Method: Non-Probability Sample
Enrollment: 488 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-12-14 (Actual); Study Completion 2025-06-14 (Estimated)

PRIMARY OUTCOMES:
Scalp-to-cortex distance will be measured using geometric brain model | Baseline
  Scalp-to-cortex distance (SCD), as a geometric feature, will measured in the Brainsight TMS neuronavigation system.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna LU, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Tai Po Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided